CLINICAL TRIAL: NCT04021316
Title: Decellularised Dermis Allograft for the Treatment of Chronic Venous Leg Ulceration
Acronym: DAVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DMC noted that the primary end point of healed index ulcer at 12 weeks was reached only in 11.5%, whereas a higher figure of 42.5% had been used for the original power calculation, suggesting the trial is significantly underpowered.
Sponsor: Imperial College London (Other)
Collaborators: University of Edinburgh (Other); Universidad de Granada (Other); University of Manchester (Other); Gloucestershire Hospitals NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); University of Birmingham (Other); NHS Blood and Transplant (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19CX5371
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Venous Ulcer; Allograft
Keywords: Compression therapy; Ulcer
MeSH Terms: conditions — Varicose Ulcer; Ulcer

STUDY DESIGN:
Intervention Model Description: Participants will undergo 1:1 web based randomisation to either standard care or the intervention via an automated system. A minimization algorithm using centre, index ulcer size and duration will be used, including a random component to lessen predictability. A separate Randomisation System Description document will contain full details of the cut-offs for index ulcer size and duration, and the probability that the allocation will be switched.
Masking Description: It is not possible to mask participants or the research/clinical teams to the treatment strategy as the DCD graft is visible after application for a period of time. However the primary outcome assessments (verification of index ulcer healing visits) will be completed by an independent clinical assessor trained in the assessment of wound healing, who will have no previous involvement with, or knowledge of, the participant's index ulcer treatment and as such will be blind to the randomised treatment strategy (as the DCD is not expected to be visible after 4 weeks).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care arm (Active Comparator): Compression bandaging therapy as per standard care
  Interventions: Other: Compression bandaging therapy
- DCD Arm (Experimental): DCD graft plus compression bandaging therapy as per standard care
  Interventions: Other: dCELL® Human Dermis (decellularised dermal skin allograft - DCD); Other: Compression bandaging therapy

INTERVENTIONS:
Other: dCELL® Human Dermis (decellularised dermal skin allograft - DCD) — DCD is produced from split thickness skin grafts (which comprise the epidermis and upper part of the dermis), and is retrieved from deceased tissue donors. All epidermal and cellular components from the dermis are removed in a patented sequential decellularisation process. As a decellularised graft, dCELL® Human Dermis fully integrates into the wound bed after application, replacing lost dermal tissue. It provides a scaffold into which the recipient's cells can grow, becoming vascularised and supporting the generation of a new epidermis, ultimately regenerating into normal skin.
  Arms: DCD Arm
Other: Compression bandaging therapy — Compression therapy will be according to local practice and may include multilayer elastic compression bandaging or stockings delivering 20 to 40mm/Hg pressure.

SUMMARY:
Does the use of decellularised dermis allograft in addition to compression therapy promote healing in chronic venous leg ulceration compared to compression therapy alone

DETAILED DESCRIPTION:
Chronic venous ulceration are open wounds on the lower limbs which have been present for at least three months and are caused by a poorly functioning venous system. The affect about 1% of the general population and about 4% of those over 65. The wounds cause pain, reduced movement, and can smell - greatly affecting the quality of life of leg ulcer patients. The standard care for these patients is compression bandaging, which requires changing several times a week by community or district nurses; this drives the high cost of leg ulcer care, which can amount to £2.5 billion per annum.

Skin grafting can be used alongside compression bandaging and can help the ulcers heal faster than compression alone. Grafts can be taken from the patient's own skin, from a donor or from tissue engineered skin. An autograft (using own skin) can cause scarring and the need for a formal surgical procedure in theatre so are not suitable for all ulcer patients. Allografts (donor skin) and xenografts (animal skin) have been used successfully, but present similar drawbacks to autografts, plus the potential for the body to reject the graft and disease transmission. Tissue engineered skin has several advantages as it has been processed to remove the cells, and therefore is won't be rejected via the immune response. Human decellularised dermis (DCD) is generated from donated skin from deceased people and processed to remove the cells. It can be glued or sewn onto the skin under local anesthetic, in an out patient setting. DCD has mainly been studied in patients with diabetic foot ulceration and has shown improved healing rates and quality of life.

This study will investigate the use of DCD in addition to compression therapy versus compression therapy alone in patients with chronic venous leg ulceration.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years or older (no upper age limit)
* The ability to consent to participation
* A diagnosis of venous leg ulceration* (defined as 'colour duplex confirmation of superficial and or deep venous reflux with any break in the skin that has either: a) been present for more than 2 weeks, or b) occurred in a person with a history of venous leg ulceration)
* Documented venous incompetence on duplex ultrasound
* Index ulcer wound duration of greater than 3 months
* Index ulcer wound size ≥ 2 cm2.
* ABPI ≥ 0.8

  * in light of the Covd-19 pandemic, the use of handheld continuous wave Dopplers will be allowed to diagnose venous disease to allow participants to be recruited from clinic without the need for an imaging appointment

Exclusion Criteria:

* A diagnosis of sickle cell
* Unable to receive one or more of the randomised treatment strategies for any reason at the discretion of the attending clinical team (e.g. known allergies to dCELL dermis preparation components)
* A clinically infected ulcer defined as evidence of erythema, cellulitis or systemically unwell
* Treatment with biomedical/topical growth factors within previous 30 days
* Previous history of an inability to tolerate compression therapy
* Foot ulcer (i.e. below the ankle)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Proportion with a healed index ulcer at 12 weeks after randomisation. | 12 weeks

SECONDARY OUTCOMES:
Time to index ulcer healing from randomisation | 12 months
The percentage change in index ulcer area in cm2 at 12 weeks from randomisation | 12 weeks
The proportion of participants with a healed index ulcer at 12 months from randomisation | 12 months
The proportion of participants whose index ulcer healed for whom an ulcer recurred at the index site within 12 months from randomisation | 12 months
Generic quality of life using the EuroQol-5D (EQ-5D) questionnaire | 12 weeks, 6 months and 12 months from randomisation
  A health index on a score of 0 to 1 and the participants' self-rated health on a vertical score of zero to 100. Higher scores indicate better quality of life
Disease specific quality of life using the Charing Cross Venous Ulcer Questionnaire (CCVUQ) | 12 weeks, 6 months and 12 months from randomisation
  Scale 0 to 100, with lower scores indicating better quality of life
The cost for each patient, calculated from the healthcare resources used | 12 months
Incremental cost-effectiveness ratio (ICER) from the EQ-5D questionnaire, with appropriate sensitivity analysis | 12 months
  An intervention may be considered cost-effective when its ICER is less than the threshold set by health policy decision-makers. In the UK, the cost-effectiveness threshold is currently in the range £20 000-30 000 per QALY

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, Principal Investigator — Imperial College London
Locations (17):
- United Kingdom (17):
  - North Bristol NHS Trust, Bristol
  - Cardiff and Vale University Health Board, Cardiff
  - North Cumbria University Hospitals NHS Trust, Carlisle
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucester
  - AT Medics, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - London North West University Healthcare, London
  - St Charles Centre for Health and Welbeing, Central London Community Healthcare NHS Trust, London
  - Aneurin Bevan University Health Board, Newport
  - Northampton General Hospital NHS Trust, Northampton
  - Livewell, Plymouth
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Swansea Bay University Health Board, Swansea
  - Taunton and Somerset NHS Foundation Trust, Taunton
  - Mid Yorkshire Hospitals NHS Trust, Wakefield
  - Worcestershire Acute Hospitals NHS Trust, Worcester

IPD SHARING:
Plan to Share IPD: No
IPD sharing will be in line with Imperial College data sharing policy